CLINICAL TRIAL: NCT07314164
Title: CaboLife: A Prospective Non-Interventional Study on Effectiveness and Safety of Cabozantinib in Real-Life Setting for Previously Treated Patients With Neuroendocrine Tumour
Brief Title: Study of Cabozantinib in Participants With Neuroendocrine Tumors Who Have Already Received Prior Treatment
Status: Recruiting | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-60000-467
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will assess how well cabozantinib works and how safe it is in adults with a type of cancer called neuroendocrine tumors (NETs).

These tumors can appear in all parts of the body. All participants in this study have already received at least one treatment that affects the whole body to help manage their cancer, but their disease has continued to grow.

The study will take place in regular hospitals and clinics in Germany and Austria.

It will follow about 150 participants who are taking cabozantinib as part of their usual care. Doctors will collect information from routine medical visits, tests, and scans to see how the cancer responds to treatment and how long participants stay on cabozantinib. They will also look at side effects and how the treatment affects participants' quality of life.

This is an observational study, which means that no extra tests or procedures will be done beyond what is normally used to care for participants with this condition.

ELIGIBILITY:
Inclusion Criteria:

Participants can join the study if they meet all of the following conditions:

* Are 18 years or older and able to give informed consent.
* Have a physician-initiated decision to start treatment with cabozantinib for neuroendocrine tumors (NETs), made before joining the study.
* Have unresectable or metastatic, well-differentiated pancreatic (pNET) or extra-pancreatic neuroendocrine tumors (epNET).
* Have already received at least one prior systemic therapy, other than somatostatin analogues.
* Have signed a written informed consent form.

Exclusion Criteria:

Participants cannot join the study if:

* They are currently participating in an interventional clinical trial, or have done so within the last 3 months before joining this study.
* They have a contraindication to cabozantinib treatment, based on the product's official prescribing information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 150 adult participants in Austria and Germany who are prescribed cabozantinib tablets for unresectable or metastatic, well differentiated extra-pancreatic (epNET) and pancreatic (pNET) neuroendocrine tumours who have progressed following at least one prior systemic therapy other than somatostatin analogues prior to entry into the study will be included.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease Control Rate (DCR) | At 6 Months
  Proportion of participants who achieve complete response, partial response, or stable disease within 6 months of cabozantinib treatment, based on radiographic assessments performed as part of routine care.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 18 Months
  Proportion of participants who achieve complete or partial response based on radiographic assessments.
Change from baseline in global and subscale scores of the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC QLQ-C30) | Baseline and Every 3 Months up to 18 Months
  A validated 30-item questionnaire designed to assess the general health-related quality of life of cancer patients. It includes: 5 functional scales (physical, role, emotional, cognitive, social), 3 symptom scales (fatigue, nausea/vomiting, pain) a global health status/QoL scale and several single items (e.g., dyspnea, insomnia, appetite loss, constipation, diarrhea, financial difficulties).
Change from baseline in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Gastrointestinal Neuroendocrine Tumors Module (EORTC QLQ-GINET21) | Baseline and Every 3 Months up to 18 Months
  A 21-item module developed to supplement the QLQ-C30 for patients with gastrointestinal neuroendocrine tumors (GI-NETs). It includes 5 scales (Endocrine symptoms, Gastrointestinal symptoms, Treatment-related side effects, Social functioning, Disease-related worries) and 5 single items (weight loss, weight gain, muscle and/or bone pain, information, sexual functioning).
Percentage of participants experiencing Adverse Events (AEs), non-serious, drug-related, or serious Adverse Events (SAEs) | Up to 18 Months
  An Adverse event (AE) is any untoward medical occurrence, temporally associated with the use of study intervention, whether or not related to the study intervention.
Percentage of participants with any dose modification due to AEs. | Up to 18 months
  Percentage of participants who experienced at least one dose reduction, interruption, or discontinuation due to adverse events during the study period.
Duration of treatment (DoT) | Up to 18 Months
  Time from first dose to last dose of cabozantinib.
Percentage of participants switching to a new line of therapy | Up to 18 Months
  Percentage of participants who initiated a new line of therapy during the study period. The type of therapy received after switch will be reported descriptively and is not considered a formal outcome measure.
Disease control rate after switch to next line of therapy | 3 Months After Therapy Switch
  Proportion of participants achieving complete response, partial response, or stable disease within 3 months after switching to a new therapy, based on radiographic assessment performed as part of routine care.
Chromogranin A Levels | Baseline and Every 3 Months up to 18 Months
  Chromogranin A blood levels measured during routine care.
Neuron-Specific Enolase blood levels. | Baseline and Every 3 Months up to 18 Months
  Neuron-Specific Enolase blood levels measured during routine care.
Time to next treatment | Up to 18 Months
  Time from first dose of cabozantinib to initiation of subsequent therapy.
Progression-Free Survival (PFS) | Up to 18 Months
  Time from first dose of cabozantinib to disease progression or death from any cause.
Progression-Free Survival Rate at 12 and 18 Months | At 12 and 18 Months
  Number of participants without disease progression or death.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (6):
- Germany (6):
  - MVZ am Klinikum Aschaffenburg, Aschaffenburg
  - MVZ fuer Haematologie und Onkologie Koeln am Sachsenring, Cologne
  - Gemeinschaftspraxis Haematologie - Onkologie, Dresden
  - Asklepios Kliniken Hamburg, Hamburg
  - MVZ Leipzig Mitte, MVZ Delitzsch, Leipzig
  - Universitaetsklinikum Wuerzburg, Würzburg

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the United States (US) and/or Europe (EU).
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/